CLINICAL TRIAL: NCT00467935
Title: A Phase I/II Study to Evaluate Scotoma Reduction in And Limited Visual Acuity in aGe Related Macular Degeneration Patients Treated With Intravitreal Lucentis
Brief Title: Scotoma Reduction in AMD Patients Treated With Ranibizumab
Acronym: SALVAGE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Retina Research Foundation (Other)
Responsible Party: Paul Beer, MD, Retina Consultants, PLLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF3933
Record Dates: First submitted 2007-04-29; First posted 2007-05-01 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Macular Degeneration
Keywords: amd; disciform; fibrosis; Lucentis; scotoma
MeSH Terms: conditions — Macular Degeneration; Glycogen Storage Disease Type II; Fibrosis; Scotoma | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: intravitreal injection Lucentis (ranibizumab) — intravitreal injection Lucentis (ranibizumab)

SUMMARY:
This is a trial aimed at patients with advanced wet macular degeneration and macular scarring treated wiht intravitreal injections of Lucentis.

DETAILED DESCRIPTION:
Patients with severe wet macular degeneration and scarring in the center of the retina may benefit from treatment if the size of the blind spot is reduced wiht injections of Lucentis.

ELIGIBILITY:
Inclusion Criteria:

* BCVA < 20/320
* Disciform macular degeneration wiht exudation

Exclusion Criteria:

* Non-amd CNV

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
scotoma reduction | 12 months

SECONDARY OUTCOMES:
improved visual function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Beer, MD, Principal Investigator — Retina Research Foundation
Locations (1):
- Retina Research Center, Slingerlands, New York, United States

REFERENCES:
- See also: Sponsor — http://www.retinaresearchfoundation.org
- See also: sponsor — http://retinaconsultants.org